CLINICAL TRIAL: NCT07198685
Title: 6 Months of Bedaquiline, Delamanid, Linezolid and Levoffoxacin in RR-TB Patients in Hubei Province
Brief Title: 6 Months of Bedaquiline(BDQ), Delamanid(DLM), Linezolid(LZD) and Levofloxacin(LFX) in RR-TB Patients in Hubei Province
Acronym: BDLL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Pulmonary Hospital (Other)
Responsible Party: Principal Investigator, Yan Hu, Shuang Wei,Vice-President, Wuhan Pulmonary Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wuhan PulmonaryH
Record Dates: First submitted 2025-07-20; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Treat to Target; Treatment Duration
Keywords: BDLL; RR/MDR-TB
MeSH Terms: interventions — bedaquiline; OPC-67683; Linezolid; Levofloxacin; Cycloserine; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group (Experimental): 6-month all-oral regimen, consisting of Bedaquiline (BDQ, B), Delamanid (DLM, D), Linezolid (LZD, L), Levofloxacin (LFX) , as known as BDLL regimen
  Interventions:
  Drug: bedaquiline Drug: delamanid Drug: linezolid Drug: Levofloxacin
  Interventions: Drug: bedaquiline; Drug: Delamanid (DLM); Drug: Linezolid (LZD); Drug: Levofloxacin
- Control group (Group A) (Active Comparator): Six months of bedaquiline, linezolid, levofloxacin, cycloserine, and clofazimine, followed by 12 months of levofloxacin, cycloserine, and clofazimine.
  Interventions: Drug: bedaquiline; Drug: Delamanid (DLM); Drug: Linezolid (LZD); Drug: Levofloxacin; Drug: Cycloserine; Drug: Clofazimine

INTERVENTIONS:
Drug: bedaquiline — Administer 400 mg orally once daily for 2 weeks, followed by 200 mg orally three times a week for 22 weeks
Drug: Delamanid (DLM) — Administer 100 mg orally, twice daily for 24 weeks.
Drug: Linezolid (LZD) — Administer 600 mg orally, once daily for 24 weeks.
Drug: Levofloxacin — test group:Administer 800 mg orally, once daily for 24 weeks;control group:Administer 800 mg orally, once daily for 72 weeks
Drug: Cycloserine — Administer 250mg orally, twice daily for 72 weeks.
  Arms: Control group (Group A)
Drug: Clofazimine — Administer 100 mg orally, once daily for 72 weeks
  Arms: Control group (Group A)

SUMMARY:
This study aims to compare the efficacy and safety of a 6-month all-oral regimen including Bedaquiline (BDQ,B), Delamanid (DLM,D), Linezolid (LZD, L), and Levofloxacin (LFX,L) to the the standard long - course treatment regimen within the Chinese population. The main questions it aims to answer are:

Is the efficacy of short regimen non-inferior to standard regimen? Is the short regimen safe enough to replace the standard regimen?

Participants will:

Be given with either short or standard regimen for RR-TB treatment Be asked to complete the scheduled visit as planned.

DETAILED DESCRIPTION:
Research Methodology:

Research Subjects: A total of 26 patients with RR - TB/MDR - TB pulmonary tuberculosis undergoing ultra - short - course treatment and 26 patients undergoing standard long - course treatment, whose conditions were confirmed by molecular biology detection techniques or tuberculosis drug susceptibility test results.

Research Methods:

1. Treatment Protocol Control Group (Group A): 6 BDQ LZD LFX CS CFZ / 12 LFX CS CFZ Experimental Group (Group B): 6 BDQ DLM LZD LFX
2. In - patient and Out - patient Treatment Both in - patient and out - patient treatments are acceptable for patients. However, it is advisable for patients to be hospitalized for a period at the beginning of treatment to ensure they can follow this treatment protocol. Hospitalization can also be arranged when adverse events occur during treatment.

Medical staff are responsible for the treatment management of patients, with the following duties:

1. Strictly manage DOT on a daily basis.
2. Ensure patients participate in all scheduled follow - up visits and examinations.
3. Closely monitor adverse events and promptly notify relevant personnel for handling.
4. Update patients' treatment cards monthly.
5. Contact patients if they fail to receive treatment as scheduled.
6. Ensure that patients currently under treatment have sufficient drug reserves for preventing adverse reactions.

Measures after Missed Doses If a patient misses a dose, the treatment course should be extended according to the number of missed days (if the consecutive missed days exceed two months, the patient will be classified as having an incomplete treatment course and withdrawn from the study as a treatment failure). However, the reasons must be recorded.

3. Baseline and During - treatment Examinations 3.1 Sputum Bacteriological Examination: Sputum smear and culture should be re - examined before treatment, monthly during the treatment process, and at 3, 6, 9, and 12 months after the completion of treatment.

3.2 Body Weight: Assess the patient's body weight before treatment and monthly. 3.3 Conduct glycated hemoglobin tests every three months. If glycated hemoglobin cannot be tested, fasting blood glucose can be used instead.

3.4 Screen for AIDS or viral hepatitis before treatment. 3.5 Detect serum creatinine monthly to screen for acute kidney injury or chronic kidney disease.

3.6 Re - examine the complete blood count before treatment and monthly. 3.7 Since linezolid is included in the treatment protocol, visual acuity tests and Ishihara tests (color - blindness tests) should be re - examined before treatment and monthly thereafter.

3.8 Electrocardiogram (ECG) should be examined before treatment and monthly during the treatment period.

3.9 Thyroid - stimulating hormone (TSH) should be detected before treatment and every three months during the treatment process.

3.10 Conduct pregnancy screening for all female patients of child - bearing age at the start of treatment.

3.11 Chest CT examinations should be performed before treatment, every three months, and at 6 - month and 12 - month follow - up periods.

3.12 Other examinations may be required as determined by the attending physician.

4. Risk Pre - plan: 4.1 Handling of Treatment Discontinuation

Some patients may discontinue the study protocol for various reasons. In such cases, patients will be evaluated by an expert panel and receive personalized treatment according to the WHO's protocol design guidelines. The most common situations include:

Drug resistance to the medications in the treatment protocol. If drug resistance to the medications in this protocol is detected, the protocol should be discontinued, and the patient should be withdrawn from the group.

Pregnancy during treatment. For pregnant patients in the first trimester, it may be recommended to modify or stop the treatment protocol and withdraw the patient from the group.

Serious adverse events. Due to severe toxic reactions, one or more medications may need to be permanently discontinued. In this case, the expert panel should carefully review the patient's medical history to determine how to modify the treatment protocol and withdraw the patient from the group.

Treatment failure. If the clinical and bacteriological responses are poor after treatment, it should be regarded as a failure. A suitable treatment protocol should be developed for the patient. Regardless of whether the protocol is changed, drug susceptibility tests should be repeated to provide information for future treatment.

4.2 Monitoring and Management of Adverse Events Patients should be screened monthly by doctors trained in the diagnosis and management of adverse events. An adverse event refers to any untoward medical occurrence in a patient or clinical research subject who is taking medications, and it does not necessarily have a causal relationship with the treatment.

The management of adverse events should consider the patient's safety and treatment needs. The medications causing adverse events may need to be suspended or the dosage reduced. For the management of adverse events caused by conventional medications, please refer to the "Companion Handbook" of the "WHO Guidelines for the Programmatic Management of Drug - Resistant Tuberculosis".

4.3 Handling of Adverse Events Adverse events should be scored according to standardized scoring tables, such as the AIDS classification table for adverse event severity ("DAIDS AE Scoring Table"), the Common Terminology Criteria for Adverse Events (CTCAE), or the MSF severity scale. All adverse events that lead to temporary or permanent discontinuation of the study treatment should be carefully managed and recorded.

Safety Reporting All serious adverse events (SAEs) that occur must be reported immediately within 72 hours. This includes events that result in death, are life - threatening, require hospitalization or an extended hospital stay (excluding non - medical reasons), cause permanent or significant disability, or lead to permanent functional abnormalities.

When an adverse event (AE) occurs, the researcher is responsible for reporting it to the principal investigator, regardless of whether it is a serious adverse event. If it is an SAE, the AE form should be filled out and reported to the PI and relevant institutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary tuberculosis that is resistant to rifampin (RIF) or to both RIF and isoniazid who initiate an all-oral treatment regimen (short or long) under routine or operational conditions will be included.
* Aged between 18 and 65 years old.
* Have never used bedaquiline, delamanid, linezolid, or levofloxacin in the past, or have used them for no more than 4 weeks.
* Positive results of mycobacterial culture (either smear-positive or smear-negative) within the recent one month, and no effective anti-tuberculosis treatment received within this one-month period; or in the absence of recent sputum culture results, smear-positive sputum and no effective anti-tuberculosis treatment administered.
* No history of respiratory failure or cardiac insufficiency, and no clinically significant arrhythmia manifestations on electrocardiogram.
* During the treatment and follow - up periods, patients are required to take medications as per the research project requirements, complete treatment monitoring, and promptly report any adverse reactions to the attending physicians.
* Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Individuals with a history of optic neuropathy or peripheral neuropathy, whom the researchers believe may experience progression/worsening during the study or are not suitable for participation in this research.
* Chronic active hepatitis, with positive results for three items: hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), and hepatitis B core antibody (anti - HBc), or HBV - DNA > 1000 CPs/mL, accompanied by elevated ALT/AST. Elevation of ALT or AST is ≥3 times the upper limit of the normal value, or elevation of total bilirubin and direct bilirubin is ≥2 times the upper limit of the normal value (if it is a temporary elevation, patients can be enrolled after recovery from treatment).
* Severe renal insufficiency (creatinine clearance rate (CrCl) less than 30 mL/min).
* Individuals who have participated in clinical trials of other unlisted new drugs within the past three months.
* Known congenital QT interval prolongation, presence of any disease that can prolong the QT interval, or a QTc > 450 ms.
* Pregnant women or women who may be pregnant.
* Any cardiac diseases capable of inducing arrhythmia, such as severe hypertension (poorly controlled blood pressure), left ventricular hypertrophy (including hypertrophic cardiomyopathy), or congestive heart failure accompanied by a reduced left ventricular ejection fraction.
* A history of known, untreated, and persistent hypothyroidism. Combined with hematogenous disseminated tuberculosis and central nervous system tuberculosis.
* A history of allergy or a known allergy to any investigational medicinal product or related substances.
* HIV-positive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
End of treatment outcome | 72 weeks after the treatment initiation
  Number of individuals experiencing each tuberculosis treatment outcome (cure, completion, death, failure, lost-to-follow-up), assessed at the end of treatment by a clinician, based on culture results

SECONDARY OUTCOMES:
The median time to Sputum Culture Conversion | Time Frame: 4-24 weeks after treatment initiation
  time from treatment initiation to the first of two consecutive negative sputum cultures without an intervening positive culture in liquid media
Final tuberculosis treatment outcome | 24, 48 and 72 weeks after treatment completion
  Number of individuals experiencing each final tuberculosis treatment outcome (cure, completion, death, failure, lost-to-follow-up, relapse), assessed at 24, 48, and 72 weeks by a clinician, based on culture results

OTHER OUTCOMES:
The frequency of grade 3 or greater adverse events among patients | 72 weeks after treatment initiation
  Assessed by a clinician based on symptomatology, subjective screening, and/or laboratory findings during treatment or follow-up. Adverse events are referenced against CTCAE 5.0.

IPD SHARING:
Plan to Share IPD: No